CLINICAL TRIAL: NCT01424722
Title: ST Monitoring to Detect ACS Events in ICD Patients
Brief Title: ST Monitoring to Detect Acute Coronary Syndrome Events in Implantable Cardioverter Defibrillator Patients
Acronym: AnalyzeST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRD_420
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: ICD Indicated patients; documented CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ST Monitoring Feature (Experimental): ST segment continous monitoring feature enabled and programmed ON
  Interventions: Device: Fortify® ST, Fortify Assura® ST, Ellipse® ST family of devices

INTERVENTIONS:
Device: Fortify® ST, Fortify Assura® ST, Ellipse® ST family of devices — Algorithm for detecting ST changes that may be indicative of an acute coronary syndrome.
  Other Names: ST Monitoring Feature

SUMMARY:
This is a prospective, non-randomized, multicenter, pivotal Investigational Device Exemption (IDE) study. The intent of this study is to demonstrate the safety and effectiveness of the ST Monitoring Feature in St Jude Medical ICD systems.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multicenter, pivotal IDE study. The intent of this study is to demonstrate the safety and effectiveness of the ST Monitoring Feature in the Fortify® ST, Fortify Assura® ST, and Ellipse® ST family of devices, as well as any future St Jude Medical devices with the same ST Monitoring Feature capabilities. Effectiveness of the device will be evaluated by analyzing the sensitivity of the ST Monitoring Feature to detect clinical events. In addition, safety of the ST Monitoring Feature will be evaluated by demonstrating a low percentage of patients with false positive events.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will meet all of the following:

  1. Have an indication for an ICD implantation or pulse generator change
  2. Have documented coronary artery disease. Documented coronary artery disease is defined as having at least one of the following present a) evidence of a prior MI on ECG and/or cardiac enzymes, b) prior revascularization (by coronary artery bypass grafting or percutaneous coronary intervention) c) angina and/or ST-T wave abnormalities indicative of ischemia on exercise stress test, nuclear stress test, or echo stress test, or d) coronary artery disease diagnosed by coronary angiography.
  3. Willing and able to comply with protocol requirements, including keeping all required visits
  4. Willing to participate in the study and able to sign an IRB approved informed consent form
  5. Be at least 18 years of age when enrolled in the study

Exclusion Criteria:

* Patients will be excluded if they meet any of the following:

  1. Are pacemaker dependent (defined as a need for ventricular pacing ≥ 20% of the time)
  2. Have NYHA Class IV Heart Failure
  3. Have persistent or permanent atrial fibrillation
  4. Have a known history of intermittent Bundle Branch Block
  5. Pregnant or planning a pregnancy during the study participation
  6. Have a life expectancy of < 1 year due to any condition
  7. Are currently participating in a clinical investigation that includes an active treatment arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2258 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gibson, MD, Principal Investigator — Boston Clinical Research Institute
Locations (96):
- United States (96):
  - Cardiovascular Associates PC, Birmingham, Alabama
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Banner Heart Hospital, Mesa, Arizona
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Carondelet Specialist Group - Southwest Heartr, Tucson, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Central Cardiology, Bakersfield, California
  - John Muir Medical Center, Concord, California
  - St. Jude Hospital, Fullerton, California
  - Cardia Care Specialists, Glendale, California
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - Long Beach Memorial, Long Beach, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - USC University Hospital, Los Angeles, California
  - Cardiac Rhythm Specialists, Inc., Northridge, California
  - Sutter Memorial Hospital, Sacramento, California
  - Colorado Cardiac Alliance, Colorado Springs, Colorado
  - Cardiology Associates of Fairfield County, Norwalk, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Cardiology Consultants PA, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Watson Clinic Center, Lakeland, Florida
  - University of Miami Hospital, Miami, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Athens Regional Medical Center, Athens, Georgia
  - Northeast Georgia Heart Center, PC, Gainesville, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northern Indiana Research Alliance, Fort Wayne, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Mid-America Cardiology Associates, PC, Kansas City, Kansas
  - Kentucky Heart Institute / King's Daughter, Ashland, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - MedStar Research Institute, Baltimore, Maryland
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - University of Massachusettts Medical Center, Worcester, Massachusetts
  - Thoracic Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Providence Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - VA Medical Center Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Lourdes Cardiology Services, Cherry Hill, New Jersey
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Southwest Heart PC, Las Cruces, New Mexico
  - Buffalo Heart Group, Buffalo, New York
  - Stony Brook Medical Center, Stony Brook, New York
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Northeast Ohio Cardiovascular Associates, Akron, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Univeristy, Columbus, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - EMH Regional Medical Center, Elyria, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oklahoma Heart Institute at Utica, Tulsa, Oklahoma
  - Capital Cardiovascular Associates, Camp Hill, Pennsylvania
  - Penn State Milton Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Columbia Cardiology Consultants, Columbia, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cardiology Consultants, Johnson City, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - St. Thomas Hospital Heart, Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Cardiology Center of Amarillo, LLP, Amarillo, Texas
  - VA Medical Center Dallas, Dallas, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - McKay-Dee Heart Services, Ogden, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Hunter Holmes McGuire VAMC, Richmond, Virginia
  - The Hope Heart Institute, Bellevue, Washington
  - The Heart Institute at Virginia Mason, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ST Monitoring Feature
Started | 2258
Completed | 0
Not Completed | 2258
Not completed — Sponsor terminated investigation | 2258

BASELINE CHARACTERISTICS:
Arm/Group | ST Monitoring Feature
Number analyzed (Participants) | 2258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1029
  >=65 years | 1229
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 424
  Male | 1834
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 41
  Native Hawaiian or Other Pacific Islander | 7
  Black or African American | 266
  White | 1899
  More than one race | 0
  Unknown or Not Reported | 34
Region of Enrollment [Number; unit: participants]
  United States | 2258

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience a False Positive ST Detection in 12 Months FU
Time Frame: 12 months
Population: The analysis population includes the number of patients with Clinical Event Committee adjudicated data related to ACS events.
Measure: Count of Participants; unit: Participants
Arm/Group | ST Monitoring Feature
Number analyzed (Participants) | 1404
Participants | 115

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected from time of implant/attempted implant though last visit for each subject (up to 5 years per subject).
Description: AEs were Observations, Complications or Other Reported Events (OREs)
  * Complications-events that required invasive intervention (reported under Serious AEs here)
  * Observations-events managed without invasive intervention (reported under Non-serious AEs here)
  * ORE-event submitted by an investigator and not associated with the investigational device, clinical study, and/or defined as an AE *Subjects may have more than 1 event in more than 1 category; # subjects in each will not add to up total
Arm/Group | ST Monitoring Feature
All-Cause Mortality (participants affected / at risk) | 270/2258
Serious Adverse Events (participants affected / at risk) | 217/2258
Other Adverse Events (participants affected / at risk) | 177/2258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST Monitoring Feature (N=2258)
Aspiration (Injury, poisoning and procedural complications) | 1 (1)
Battery Depletion at Implant (Product Issues) | 1 (1)
Bleeding (Injury, poisoning and procedural complications) | 3 (3)
Cardiac Perforation (Injury, poisoning and procedural complications) | 5 (5)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 2 (2)
Cardiac/respiratory arrest (Injury, poisoning and procedural complications) | 2 (2)
Coronary sinus perforation/dissection (Injury, poisoning and procedural complications) | 1 (1)
Decompensated Heart Failure (Injury, poisoning and procedural complications) | 2 (2)
Device infection/erosion (Infections and infestations) | 24 (27)
Device Malfunction (Product Issues) | 11 (11)
Discomfort at implant site (Injury, poisoning and procedural complications) | 6 (7)
Elevated pacing thresholds (Product Issues) | 7 (7)
Endocarditis (Cardiac disorders) | 8 (8)
Generator changeout/upgrade (Product Issues) | 1 (1)
Genitourinary disease/disorder (Renal and urinary disorders) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 8 (8)
High Defibrillation Threshold (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Injury, poisoning and procedural complications) | 4 (4)
Inappropriate therapy due to non-ventricular rhythm (Product Issues) | 10 (13)
Infection (Infections and infestations) | 10 (10)
Lead dislodgment or migration (Product Issues) | 62 (68)
Lead entanglement (Injury, poisoning and procedural complications) | 1 (1)
Lead fracture (Product Issues) | 13 (13)
Lead Impedance out of range (Product Issues) | 13 (13)
Lead insulation damage (Product Issues) | 2 (2)
Lead noise (Product Issues) | 3 (4)
Loss of capture (Product Issues) | 5 (5)
Oversensing (Product Issues) | 2 (2)
pericardial effusion (Injury, poisoning and procedural complications) | 1 (1)
Pericarditis (Injury, poisoning and procedural complications) | 2 (3)
Pneumothorax (Injury, poisoning and procedural complications) | 8 (8)
Sepsis (Infections and infestations) | 4 (4)
Thrombus (Blood and lymphatic system disorders) | 1 (1)
Undersensing (Product Issues) | 2 (2)
Upper extremity thromboembolism (Blood and lymphatic system disorders) | 4 (4)
Vascular Injury/Repair (Injury, poisoning and procedural complications) | 2 (2)
Inappropriate therapy due to oversensing (Product Issues) | 4 (4)
Lead abrasion (Product Issues) | 1 (1)
Premature battery depletion (Product Issues) | 2 (2)
Vascular disease/disorder (Vascular disorders) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ST Monitoring Feature (N=2258)
Atrial Arrhythmia (Cardiac disorders) | 1 (1)
Bleeding (Injury, poisoning and procedural complications) | 7 (7)
Fluid accumulation (Injury, poisoning and procedural complications) | 1 (1)
Hypertension/hypertensive crisis (Vascular disorders) | 1 (1)
Inappropriate therapy due to non-ventricular rhythm (Product Issues) | 46 (50)
Infection (Infections and infestations) | 7 (7)
Lead Fracture (Product Issues) | 3 (3)
Lead noise (Product Issues) | 1 (1)
Pacemaker mediated tachycardia (Product Issues) | 10 (11)
Stroke/Cerebrovascular accident (Nervous system disorders) | 3 (3)
Thrombus (Blood and lymphatic system disorders) | 3 (3)
Ventricular Arrhythmia (Cardiac disorders) | 2 (2)
Allergic reaction (Injury, poisoning and procedural complications) | 3 (3)
Cardiac perforation (Injury, poisoning and procedural complications) | 1 (1)
Chest pain - non cardiac (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive changes (Injury, poisoning and procedural complications) | 1 (1)
Device infection/erosion (Infections and infestations) | 2 (2)
Device malfunction (Product Issues) | 5 (5)
Discomfort at incision/implant site (Injury, poisoning and procedural complications) | 9 (10)
Edema (Injury, poisoning and procedural complications) | 1 (1)
Exercise limitation (General disorders) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 24 (24)
Inappropriate therapy due to oversensing (Product Issues) | 6 (6)
Lead impedance out of range (Product Issues) | 9 (10)
Lead insulation damage (Product Issues) | 2 (2)
Loss of capture (Product Issues) | 2 (2)
Musculoskeletal disease/disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-SJM hardware related problem (Product Issues) | 1 (1)
Oversensing (Product Issues) | 5 (5)
Pericardial effusion (Injury, poisoning and procedural complications) | 2 (2)
Pericarditis (Injury, poisoning and procedural complications) | 2 (2)
Phantom shock (Psychiatric disorders) | 2 (2) — Subject imagined shock from device
Pneumothorax (Injury, poisoning and procedural complications) | 4 (4)
Possible generator migration (Product Issues) | 1 (1)
Skin disease/disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)
Suture protrusion (Injury, poisoning and procedural complications) | 1 (1)
Syncope/pre-syncope (General disorders) | 2 (2)
Undersensing (Product Issues) | 2 (2)
Upper extremity thromboembolism (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Statistical Analysis Plan (2013-02-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT01424722/SAP_000.pdf
  • Study Protocol (2013-02-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT01424722/Prot_001.pdf
  • Informed Consent Form (2013-06-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT01424722/ICF_002.pdf